CLINICAL TRIAL: NCT04765631
Title: Type 2 Diabetes and Bone Microarchitecture in Men and Women: a Case-control Study
Brief Title: Type 2 Diabetes and Bone Microarchitecture
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Type 2 diabetes bone
Record Dates: First submitted 2020-07-23; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Type 2 diabetes: Subjects from 3 cohorts (QUALYOR, OFELY, STRAMBO) presenting type 2 diabetes
  Interventions: Other: Patients with Type 2 diabetes
- Control subjects without Type 2 diabetes: Controls patients from 3 cohorts (QUALYOR, OFELY, STRAMBO) without type 2 diabetes
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Patients with Type 2 diabetes — No intervention
  Groups: Patients with Type 2 diabetes
Other: Placebo — Placebo comparator
  Groups: Control subjects without Type 2 diabetes

SUMMARY:
Type 2 diabetes is a major public health problem, associated with an increased risk of fractures. Diabetes even appears to be the most important predictor of low kinetic fractures in men and women, and the risk of hip fracture in type 2 diabetics is increased by 40 to 50%, with often more serious consequences (post-operative complications, longer hospital stays, increased mortality rate).

Currently, the risk of fractures is estimated by the measure of areal bone mineral density (aBMD) and T-score. However, in diabetics aBMD is not decreased, and even paradoxically increased. Indeed, aBMD is 5-10% higher in type 2 diabetic patients compared to non-diabetic subjects, which suggests that the assessment of fracture risk in these patients is underestimated. The High Resolution peripheral Quantitative Computed Tomography (HR-pQCT) 3D bone imaging technique has a resolution close to the size of the bone trabeculae. It is used to assess volumetric bone mineral density (vBMD) and bone microarchitecture at the tibia and distal radius, and enables a better estimation of the fracture risk compared to the measurement of aBMD. Our hypothesis is that bone microarchitecture is altered in type 2 diabetic patients, explaining the increased risk of fracture in this population compared to non-diabetics.

We propose to set up a descriptive case control study, nestled in 3 cohorts of men and women (QUALYOR, OFELY and STRAMBO), to compare the bone micro-architecture measured by HR-pQCT at the level of the tibia and distal radius, in type 2 diabetics compared to non-diabetic subjects from the same cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Men and women included in the 3 cohorts (QUALYOR, OFELY, STRAMBO) presenting type 2 diabetes
* Age- and sex-matched control patients from the same cohorts without type 2 diabetes ; two control were age- and sex-matched to one type 2 diabetes patient.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women included in the 3 cohorts (QUALYOR, OFELY, STRAMBO)
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
The main outcome is the comparison of total volumetric bone mineral density (vBMD) at the tibia and distal radius, in type 2 diabetics compared to non-diabetic subjects. | at inclusion for Qualyor patients. (the HRpQCT measure considered in this study is realised at the first visit just after inclusion of the patient for the Qualyor patients)
  The main outcome is the comparison of total volumetric bone mineral density (vBMD) measured by HR-pQCT at the tibia and distal radius, in type 2 diabetics compared to non-diabetic subjects from 3 cohorts of men and women (QUALYOR, OFELY, STRAMBO).

CONTACTS AND LOCATIONS:
Locations (1):
- INSERM U1033, pavillon F, Hôpital E. Herriot. 5, place d'Arsonval, Lyon, France